CLINICAL TRIAL: NCT00005697
Title: Intervention for Resistant Pregnant Smokers
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4272; R01HL050815 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
This 31-month supplement to Sustaining Women's Smoking Cessation Postpartum (Project PANDA) designed, implemented, and evaluated an intensified intervention for pregnant women who were unable to stop smoking with minimal assistance.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The substudy was a population-based experiment with White, Black, and Hispanic pregnant women whose continued smoking made them ineligible for randomization into the parent study. It was unique in focusing on heavier, more addicted pregnant smokers. PANDA research sites and protocols offered a special opportunity for a low cost test of a disseminable intervention which this project team was uniquely qualified to design and implement. The new intervention, One- to-One, used telephone counselors to assess the counselee's stage in the change process and give stage-appropriate messages, using established techniques of motivational interviewing. Between the two counselor calls spaced 10 days apart, counselees received personalized written feedback and suggestions. The primary aim, increasing quitting during pregnancy, was assessed by unobtrusive urine samples taken during prenatal visits in the ninth month and identified only by study group.

A series of postpartum interviews with subsample cotinine validation was used to examine the second important aim, reduction of infant smoke exposure. A combination of messages, peer modeling, and support helped women sustain cessation after delivery and eliminate smoking around the baby. Project PANDA videotapes and newsletters already contained these messages and required only minimal supplementation to be used with the One-to-One experimental group, regardless of their success in quitting in pregnancy. As in Project PANDA, the assessments were separated from the experiment by enrolling subjects in a university-sponsored study of new mothers' health practices and baby care and by presenting the program as usual care by the health care site.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01; Study Completion 1996-12

REFERENCES:
- [Background] Hudmon KS, Mullen PD, Nicol L, Hammond SK, Sockrider MM, Sajak T, Thompson J. Telephone-guided placement and removal of nicotine monitors for the assessment of passive exposure to environmental tobacco smoke. Toxicol Ind Health. 1997 Jan-Feb;13(1):73-80. doi: 10.1177/074823379701300107. PMID 9098952
- [Background] Mullen PD, Pollak KI, Titus JP, Sockrider MM, Moy JG. Prenatal smoking cessation counseling by Texas obstetricians. Birth. 1998 Mar;25(1):25-31. doi: 10.1046/j.1523-536x.1998.00025.x. PMID 9534502
- [Background] Groff JY, Mullen PD, Mongoven M, Burau K. Prenatal weight gain patterns and infant birthweight associated with maternal smoking. Birth. 1997 Dec;24(4):234-9. doi: 10.1111/j.1523-536x.1997.tb00596.x. PMID 9460314
- [Background] Mongoven M, Dolan-Mullen P, Groff JY, Nicol L, Burau K. Weight gain associated with prenatal smoking cessation in white, non-Hispanic women. Am J Obstet Gynecol. 1996 Jan;174(1 Pt 1):72-7. doi: 10.1016/s0002-9378(96)70376-9. PMID 8572037